CLINICAL TRIAL: NCT06792253
Title: Phase Ⅲ Clinical Trial Comparing BEBT-908 Combined With Rituximab (R) to Standard of Care for the Treatment of Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Study Comparing BEBT-908 Combined With R to SOC for the Treatment of Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-908-P08
Record Dates: First submitted 2025-01-16; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Keywords: BEBT-908; Efficacy; Safety
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Injections; BEBT-908; Rituximab; Gemcitabine; Oxaliplatin; Etoposide; Ifosfamide; Carboplatin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned in a 1:1 ratio to either the experimental group (BEBT-908 combined with R) or the control group [investigator-selected standard chemotherapy regimen (R-GemOx or R-ICE)].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (BEBT-908 Combined With R) (Experimental): Ifupinostat Hydrochloride for Injection,18.5mg/m^2 each time,is administered on days 1, 3, 5, 8, 10, and 12 of each cycle during cycles 1 to 8,with a 21-day cycle duration. After cycle 8, participants without PD enter a maintenance treatment phase that can last up to 24 months: Medication is administered on days 1, 3, 5, 8, 10, and 12 of each cycle, with a 21-day cycle duration, or as assessed by the investigator, medication is administered on days 1, 3, 5, 8, 10, and 12 of each cycle, with a 42-day cycle duration.
  Rituximab Injection,375 mg/m^2 each time,is administered on day 1 of each cycle during cycles 1 to 8. After cycle 8, medication is administered on day 1 of every third cycle, with a 21-day cycle duration.
  Interventions: Drug: Ifupinostat Hydrochloride for Injection; Drug: Rituximab Injection
- Control Group (R-GemOx or R-ICE) (Active Comparator): Rituximab Injection,375mg/m^2 each time,is administered on day 1 of each cycle,with a 21-day cycle duration, for a total of 8 treatment cycles.
  Gemcitabine Hydrochloride for Injection,1g/m^2 each time,is administered on day 2 of each cycle,with a 21-day cycle duration, for a total of 8 treatment cycles.
  Oxaliplatin Injection,100mg/m^2 each time,is administered on day 2 of each cycle, with a 21-day cycle duration, for a total of 8 treatment cycles.
  Etoposide Injection,100mg/m^2 each time,is administered on days 1, 2, and 3 of each cycle, with a 21-day cycle duration, for a total of 8 treatment cycles.
  Ifosfamide for Injection,5000mg/m^2 each time,is administered on day 2 of each cycle, with a 21-day cycle duration, for a total of 8 treatment cycles.
  Carboplatin Injection, with a single dose ≤800 mg [calculated based on area under the curve(AUC)=5],is administered on day 2 of each cycle, with a 21-day cycle duration, for a total of 8 treatment cycles.
  Interventions: Drug: Rituximab Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Oxaliplatin Injection; Drug: Etoposide Injection; Drug: Ifosfamide for Injection; Drug: Carboplatin Injection

INTERVENTIONS:
Drug: Ifupinostat Hydrochloride for Injection — Ifupinostat Hydrochloride for Injection,dosage of administration:18.5mg/m^2,frequency and duration of administration:Medication is administered on days 1, 3, 5, 8, 10, and 12 of each cycle,with a 21-day or 42-day cycle duration.
  Other Names: BEBT-908 for Injection; CUDC-908
  Arms: Experimental Group (BEBT-908 Combined With R)
Drug: Rituximab Injection — Rituximab Injection,dosage of administration:375 mg/m^2,frequency and duration of administration:Medication is administered on day 1 of each cycle or every third cycle, with a 21-day cycle duration.
  Other Names: IDEC-C2B8
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine Hydrochloride for Injection,dosage of administration:1g/m^2,frequency and duration of administration:Medication is administered on day 2 of each cycle, with a 21-day cycle duration.
  Other Names: NSC 613327
  Arms: Control Group (R-GemOx or R-ICE)
Drug: Oxaliplatin Injection — Oxaliplatin Injection,dosage of administration:100mg/m^2,frequency and duration of administration:Medication is administered on day 2 of each cycle, with a 21-day cycle duration.
  Other Names: NSC 266046
  Arms: Control Group (R-GemOx or R-ICE)
Drug: Etoposide Injection — Etoposide Injection,dosage of administration:100mg/m^2,frequency and duration of administration:Medication is administered on days 1,2,and 3 of each cycle, with a 21-day cycle duration.
  Other Names: VP-16213
  Arms: Control Group (R-GemOx or R-ICE)
Drug: Ifosfamide for Injection — Ifosfamide for Injection,dosage of administration:5000mg/m^2,frequency and duration of administration:Medication is administered on day 2 of each cycle, with a 21-day cycle duration.
  Other Names: NSC109724
  Arms: Control Group (R-GemOx or R-ICE)
Drug: Carboplatin Injection — Carboplatin Injection,,dosage of administration:single dose ≤800 mg (calculated based on AUC=5),frequency and duration of administration:Medication is administered on day 2 of each cycle, with a 21-day cycle duration.
  Other Names: NSC 241240
  Arms: Control Group (R-GemOx or R-ICE)

SUMMARY:
This is a multicenter, randomized, controlled, open-label Phase III clinical trial, aimed at evaluating the efficacy and safety of BEBT-908 combined with rituximab (R) compared to investigator-selected standard chemotherapy regimens [Standard of Care (SOC)] [i.e., rituximab-gemcitabine-oxaliplatin (R-GemOx) or rituximab-ifosfamide-carboplatin-etoposide (R-ICE)] for the treatment of relapsed/refractory diffuse large B-cell lymphoma (r/r DLBCL).

DETAILED DESCRIPTION:
The study will recruit 416 subjects, who will be randomly assigned in a 1:1 ratio to either the experimental group (BEBT-908 combined with R) or the control group [investigator-selected standard chemotherapy regimen (R-GemOx or R-ICE)]. Approximately 208 subjects will be enrolled in the experimental group, and approximately 208 in the control group. The treatment cycle is 21 days, with a total of 8 treatment cycles. The experimental group will receive BEBT-908 + R treatment from cycles 1 to 8; participants who do not appear progressive disease (PD) after cycle 8 may continue to receive BEBT-908 and/or R treatment, entering a maintenance phase of up to 24 months. The control group will receive the investigator-selected SOC (i.e., R-GemOx or R-ICE) treatment from cycles 1 to 8, and will not receive further study medication after cycle 8.

Each subject's study process includes three phases: screening, treatment, and post-treatment follow-up. The screening phase can last up to 21 days. During the treatment phase, tumor assessments will be conducted every 6 weeks (±7 days) within the first 8 treatment cycles, and every 9 weeks (±7 days) after cycle 8.After the end of treatment, safety follow-up will be conducted on day 28 (+7 days) after the last dose, efficacy follow-up will be conducted every 9 weeks (±7 days), and survival follow-up will be conducted every 3 months (±2 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. The subject has been fully informed and is willing to sign the Informed Consent Form (ICF).
2. Age is ≥18 years and ≤75 years, both men and women are eligible.
3. Pathologically diagnosed as diffuse large B-cell lymphoma according to the 2022 World Health Organization classification, confirmed by central pathology review (Patients who relapse after more than one year need to undergo tissue biopsy again to confirm the pathological diagnosis.).
4. Measurable lesions [The criteria for measurable lesions are: the longest diameter of lymph node lesions measured by enhanced Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) is greater than 15 mm, and the longest diameter of extranodal lesions is greater than 10 mm.] assessed by Positron Emission Tomography/Computed Tomography (PET-CT) and Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) according to the Lugano 2014 criteria .
5. Must have relapsed or refractory diffuse large B-cell lymphoma after at least one systemic therapy [Salvage chemotherapy and immunotherapy after stem cell transplantation will be considered as first-line systemic treatment; maintenance therapy will not be counted as a separate line of systemic treatment; local radiotherapy for diffuse large B-cell lymphoma (DLBCL) aimed at cure will not be counted as first-line systemic treatment; patients who do not achieve PR after four cycles of first-line treatment are eligible for the study; patients who do not achieve PR after two cycles of second-line or higher treatment are eligible for the study. Primary refractory DLBCL patients are defined as those who have no response during first-line treatment or relapse within six months after the end of treatment, and they will be allowed to participate in the study. Patients who relapse within 12 months after stem cell transplantation are also eligible for inclusion. Refractory DLBCL patients are those who do not achieve response after adequate front-line treatment (at least four cycles of first-line chemotherapy, or at least two cycles of subsequent treatment), or who progress during previous first-line treatment, or who progress within six months (less than six months) after achieving response to previous adequate front-line treatment, or who relapse within 12 months after achieving response to stem cell transplantation. Relapsed DLBCL patients are those who relapse six months or more after achieving response to previous adequate front-line treatment, or who relapse 12 months or more after achieving response to stem cell transplantation.], and at least one systemic therapy must include CD20 antibody.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
7. Expected survival >12 weeks.
8. Organ function levels must meet the following requirements:

Peripheral blood:

1. Absolute neutrophil count (ANC) ≥1.0×10^9/L;
2. Hemoglobin (HGB) ≥80g/L;
3. Platelet count (PLT) ≥100×10^9/L;

Liver and kidney function:

1. Serum total bilirubin ≤1.5×Upper Limit of Normal (ULN) (for patients with Gilbert syndrome, total bilirubin <3.0×ULN with direct bilirubin within normal range);
2. Serum creatinine <1.5×ULN;
3. Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) ≤2.5×ULN (≤5×ULN if there is liver involvement).

Exclusion Criteria:

1. Known severe allergy to the study drug or any of its excipients;
2. Due to the potential genotoxicity, mutagenicity, and teratogenicity of the study drug, the following subjects should be excluded:

   1. Men and women who have not undergone in vitro preservation of sperm or oocytes and plan to have children within 5 years, unless subsequent studies confirm reproductive safety;
   2. Pregnant or breastfeeding women;
3. Primary central nervous system lymphoma;
4. DLBCL with active central nervous system brain metastases or meningeal involvement at the time of screening;
5. Other active malignant tumors that require treatment and may interfere with the study.
6. Treatment history before the trial:

   1. Received other small molecule targeted drug therapy within 2 weeks before enrollment;
   2. Previously received BEBT-908 or R-ICE and R-GemOx therapy before enrollment;
   3. Underwent autologous hematopoietic stem cell transplantation within 3 months before enrollment;
   4. Received radiotherapy that affects the evaluation of the efficacy of this study within 3 months before enrollment, or local supportive radiotherapy that affects the subject's bone marrow function;
   5. Underwent myelosuppressive chemotherapy or biological therapy within 3 weeks before enrollment;
   6. Used traditional Chinese medicine and patent medicine with antitumor effects within 2 weeks before enrollment;
   7. Underwent major surgery (Referring to the Level 3 and Level 4 surgeries as stipulated in the "Administrative Measures for the Clinical Application of Medical Technologies" implemented on May 1, 2009.) other than tumor biopsy within 4 weeks before enrollment, or the side effects of the surgery have not yet stabilized;
   8. Received any hematopoietic cell colony-stimulating factor therapy (such as granulocyte colony-stimulating factor G-CSF, granulocyte-macrophage colony-stimulating factor GM-CSF) or thrombopoietin TPO therapy (Subjects who have started receiving erythropoiesis-stimulating agents or darbepoetin within 2 weeks prior to enrollment are eligible for inclusion.) within 2 weeks before enrollment;
   9. Received prednisone >10mg per day (or other equivalent doses of glucocorticoids) within 7 days before enrollment [If used for the treatment of diseases other than lymphoma, such as rheumatoid arthritis, polymyalgia rheumatica, adrenal insufficiency, or asthma, subjects may receive a stable dose of up to 10 mg per day of prednisone (or an equivalent dose of other glucocorticoids).];
   10. Underwent chimeric antigen receptor T cell immunotherapy (CAR-T therapy) within 3 months before enrollment.
7. After the previous treatment (chemotherapy or biological therapy), there are persistent Grade 2 or higher [Common Terminology Criteria for Adverse Events (CTCAE) V5.0 criteria] toxicities that have not stabilized at the time of enrollment (alopecia excluded);
8. There is an active clinical severe infection of Grade 2 or higher (CTCAE V5.0 criteria);
9. Co-morbid conditions:

   1. Poorly controlled diabetes mellitus [with a random blood glucose level ≥11.1 mmol/L or Glycosylated Hemoglobin, Type A1C (HbA1c) ≥8.5% despite hypoglycemic treatment];
   2. Severe pulmonary disease (CTCAE V5.0 Grade III-IV);
   3. Severe cardiac disease [Including any of the following: left ventricular ejection fraction (LVEF) <50% detected by cardiac radionuclide scan [Multigated Acquisition (MUGA)] or echocardiogram (ECHO); Fridericia-corrected QT value (QTcF interval) >450ms for males and > 470ms for females (QTcF formula); unstable angina; symptomatic pericarditis; myocardial infarction within the past 6 months with persistent elevation of cardiac enzymes or persistent regional left ventricular wall abnormalities recorded during LVEF measurement; history of congestive heart failure (New York Heart Association Class III-IV), or history of cardiomyopathy.].
   4. Significant renal or hepatic dysfunction;
   5. Uncontrolled active hepatitis B, hepatitis C, syphilis (individuals with both specific and non-specific syphilis antibodies positive), and active Epstein-Barr virus infection [The following active infections with clinical significance, including hepatitis B (HBV), hepatitis C (HCV), and syphilis. Active hepatitis B is defined as: hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg) or hepatitis B core antibody positive, and HBV DNA ≥ 2000 IU/ml (approximately equal to 10^4 copies/ml), hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg) positive, HBV DNA < 2000 IU/ml, according to the requirements of infectious disease control, the subject should continue to take antiviral drug treatment); active hepatitis C is defined as: HCV RNA above the upper limit of detection; positive syphilis spirochete antibody test, should be tested for non-specific syphilis spirochete antibodies [Rapid Plasma Reagin Test (PRP) or Toluidine Red Unheated Serum Test (TRUST)], the latter is negative and the subject is judged by the researcher to have been infected with syphilis in the past but has been cured can be included; current EB virus infection refers to EB virus serological detection of Epstein-Barr Virus Capsid Antigen Immunoglobulin M (VCA-IgM), Epstein-Barr Virus Early Antigen Immunoglobulin G (EA-IgG) positive or EB virus DNA test positive.];
   6. Known positive for human immunodeficiency virus (HIV);
   7. History of mental illness, family history of mental illness, or mood disorders as judged by the investigator or psychiatrist [Including a medical history of depressive episodes, bipolar disorder (Type I or II), obsessive-compulsive disorder, schizophrenia, suicide attempts or suicidal ideation, or thoughts of killing (immediate risk of harming others), and anxiety levels above Grade 3.], and deemed unsuitable for enrollment by the investigator;
   8. Need for concomitant anticoagulant or antiplatelet therapy during the study period;
   9. Uncontrolled hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg);
   10. Severe internal medical conditions with a risk of major bleeding or a history of major bleeding.
10. Concurrent use of drugs that may cause QT interval prolongation or torsades de pointes;
11. Within 4 weeks prior to enrollment, currently receiving or requiring treatment with strong inhibitors or inducers of cytochrome P450 (CYP) 3A4 isoenzyme after enrollment (Within 4 weeks prior to enrollment and during the study period, subjects must not receive treatment with strong inhibitors or inducers of the cytochrome P450 (CYP) 3A4 isoenzyme. However, concurrent treatment with moderate or weak CYP3A4 inhibitors is permitted.);
12. Within 4 weeks prior to enrollment, participated in other clinical trials and used investigational drugs;
13. Any unstable condition or situation that may jeopardize the subject's safety and compliance with the study as judged by the investigator;
14. Subjects deemed unsuitable for treatment with this protocol by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 48 months
  Defined as the time from the date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 48 months
  Defined as the time from randomization to tumor progression or death, whichever occurs first.
Overall Response Rate (ORR) | Up to 48 months
  Defined as the proportion of subjects achieving complete response (CR) and partial response (PR) from the start of randomization to tumor progression among the total number of subjects.
Overall Response Rate After Completion of Treatment (ORR-EoT) | Up to 8 treatment cycles (Each cycle is 21 days.)
  Defined as the proportion of subjects achieving complete response (CR) and partial response (PR) after the subject has completed eight cycles of treatment among the total number of subjects.
Clinical Benefit Rate (CBR) | Up to 48 months
  Defined as the percentage of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) from the start of randomization to the time of tumor progression.
Duration of Response (DoR) | Up to 48 months
  Defined as the time interval from the first assessment of complete response (CR) or partial response (PR) to the occurrence of progressive disease (PD) or death due to any cause.
Occurrence of Adverse Events (AEs) | Up to 48 months
  Occurrence of AEs will be graded according to the revised National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE V5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Phd, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China